CLINICAL TRIAL: NCT00733707
Title: Improving Adherence With Oral Contraceptives Using Daily Text Messaging Reminders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Grant-806
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Oral Contraceptive Pill Adherence
Keywords: adherence; oral contraceptive pills; contraception; text messaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Text messaging reminders
  Interventions: Behavioral: Text messaging reminders
- 2 (No Intervention): No text messaging reminder

INTERVENTIONS:
Behavioral: Text messaging reminders — Subjects in this arm will receive daily text message reminders once per day at the same time each day. Messages will remind the subject to take their oral contraceptive pill.
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether there is increased oral contraceptive pill (OCP) adherence in women receiving daily text messaging reminders to take their OCP, compared to women who do not receive reminders. The investigators hypothesize that women who receive daily text messaging reminders to take their OCP will have increased pill adherence compared to women who do not receive reminders.

The investigators also hope to determine whether there is a difference in OCP adherence as measured by electronic monitoring device and wireless real-time data collection versus traditional patient pill diaries. The investigators hypothesize that electronic monitoring device and wireless real-time data collection will demonstrate lower adherence compared to traditional patient pill diaries.

ELIGIBILITY:
Inclusion Criteria:

* Using oral contraceptive pills (OCPs) for less than 1 month, or plan to initiate OCP use at their current visit
* Be willing to use OCPs that are on formulary for the duration of the study
* Having a personal mobile phone with text messaging capabilities
* Proficiency in English or Spanish
* Agreeing to surveys regarding demographics, pill adherence behavior and its influences
* If younger than 18, must be accompanied by a parent or legal guardian who can provide informed consent for research participation

Exclusion Criteria:

* Electing OCPs solely for non-contraceptive benefits only
* Interest in pregnancy within the next 12 months
* Inability to give informed consent
* Planning to move from the local area before study completion, and is unable to return for follow-up and return the electronic pill bottle
* Planning travel outside the cell phone networks of United States or Canada
* Being in a situation where receiving text messages to take a birth control pill may endanger the safety of the subject

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Average number of missed pills per cycle | 3 months

SECONDARY OUTCOMES:
Rate of adherence as recorded by the electronic pill-dispensing device versus the rate of adherence as recorded by patient pill diaries | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jane Doe, Principal Investigator — Planned Parenthood
Locations (1):
- Planned Parenthood League of Massachusetts, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hou MY, Hurwitz S, Kavanagh E, Fortin J, Goldberg AB. Using daily text-message reminders to improve adherence with oral contraceptives: a randomized controlled trial. Obstet Gynecol. 2010 Sep;116(3):633-640. doi: 10.1097/AOG.0b013e3181eb6b0f. PMID 20733446